CLINICAL TRIAL: NCT07208461
Title: A Phase Ⅱ, Randomized, Observer-blinded, Placebo-Controlled Clinical Trial to Assess the Immunogenicity and Safety of the Respiratory Syncytial Virus (RSV) Vaccine, LYB005 in Older Adults Aged 60 Years and Older
Brief Title: A Study to Evaluate the Immunogenicity and Safety of a Recombinant Respiratory Syncytial Virus Vaccine in Older Adults Aged 60 Years and Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LYB005/CT-CHN-201
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infection Prevention
Keywords: Respiratory Syncytial Virus; Respiratory Syncytial Virus Infection; Recombinant Respiratory Syncytial Virus (RSV) Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Low dose antigen of LYB005 without A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (low dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: Low dose antigen of LYB005 without A01B adjuvant
- Low dose antigen of LYB005 with A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (low dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: Low dose antigen of LYB005 with A01B adjuvant
- Middle dose antigen of LYB005 without A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (middle dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: Middle dose antigen of LYB005 without A01B adjuvant
- Middle dose antigen of LYB005 with A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (middle dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: Middle dose antigen of LYB005 with A01B adjuvant
- High dose antigen of LYB005 without A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (high dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: High dose antigen of LYB005 without A01B adjuvant
- High dose antigen of LYB005 with A01B adjuvant (Experimental): Participant aged 60 years and older will be vaccinated with 1 dose of LYB005 (high dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: High dose antigen of LYB005 with A01B adjuvant
- Placebo (Placebo Comparator): Participants aged 60 years and older will be vaccinated with 1 dose of placebo at Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 30 μg antigen without A01B adjuvant.
  Arms: Low dose antigen of LYB005 without A01B adjuvant
Biological: Low dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 30 μg antigen adjuvanted with A01B.
  Arms: Low dose antigen of LYB005 with A01B adjuvant
Biological: Middle dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 60 μg antigen without A01B adjuvant.
  Arms: Middle dose antigen of LYB005 without A01B adjuvant
Biological: Middle dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 60 μg antigen adjuvanted with A01B.
  Arms: Middle dose antigen of LYB005 with A01B adjuvant
Biological: High dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 120 μg antigen without A01B adjuvant.
  Arms: High dose antigen of LYB005 without A01B adjuvant
Biological: High dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 120 μg antigen adjuvanted with A01B.
  Arms: High dose antigen of LYB005 with A01B adjuvant
Biological: Placebo — 0.5 mL 0.9% sodium chloride (normal saline) injection per dose
  Arms: Placebo

SUMMARY:
This is a randomized, observer-blinded, placebo-controlled Phase Ⅱ clinical trial to evaluate the immunogenicity and safety of the Respiratory Syncytial Virus (RSV) Vaccine, LYB005 in participants aged 60 years and older.

DETAILED DESCRIPTION:
A randomized, observer-blinded, placebo-controlled trial will be conducted to observe the immunogenicity and safety of LYB005 in adults aged 60 years and older. A total of 700 participants aged 60 years and older will be enrolled. Six formulations of LYB005 will be provided, three dose levels of antigen with or without A01B adjuvant. All participants will randomly receive six investigational vaccines and the placebo in a 1:1:1:1:1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Residents aged 60 years and older (at the time of screening), regardless of gender;
2. Participants can provide valid identification, voluntarily agree to participate in the study, and sign the Informed Consent Form, and are able to attend all planned follow-up visits and comply with the protocol requirements;
3. Axillary temperature < 37.3°C on the day of enrollment;
4. Female participants must be postmenopausal (postmenopausal status defined as amenorrhea for 12 months without other medical causes) and must not intend to become pregnant by any means. Male participants must practice strict contraception and avoid plans for procreation or sperm donation from the screening period until 1 month after vaccination. Acceptable methods of contraception include oral contraceptives (excluding emergency contraception), injectable or implantable contraception, sustained-release local contraceptives, contraceptive patches, intrauterine devices, sterilization, abstinence, condoms, diaphragms, and cervical caps.

Exclusion Criteria:

1. Allergy to the investigational vaccine or its excipients, or a history of anaphylactic shock or other serious adverse reactions to other vaccines;
2. Previous vaccination against Respiratory Syncytial Virus;
3. A confirmed diagnosis or etiological evidence of respiratory syncytial virus infection and related diseases caused by the infection within 12 months before enrollment;
4. Has taken antipyretics, analgesics or anti-allergy drugs within 24 hours before enrollment;
5. Has received any vaccine within 14 days before vaccination, or have received a live vaccine within 28 days;
6. Has received blood or blood-related products, including immunoglobulin, within 3 months prior to enrollment; or plan to use them during the study period;
7. Individual with the following diseases: ①Has acute diseases or are in the acute exacerbation period of chronic diseases within 3 days before vaccination; ②Diagnosed with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.; ③History of congenital or acquired immunodeficiency or autoimmune diseases; Chronic administration (≥14 consecutive days) of corticosteroids (dose ≥ 20 mg/day prednisone or equivalent dose) or other immunosuppressants within the past 3 months, with the exception of inhaled or topical steroids, or short-term use (<14 consecutive days) of oral corticosteroids; ④Neurological diseases or family history (seizures, epilepsy, encephalopathy, etc.); history of psychiatric disorders or family history; ⑤Asplenia or functional asplenia; ⑥Severe or uncontrolled or hospitalization-required cardiovascular diseases, diabetes, blood and lymphatic system diseases, immune system diseases, liver and kidney diseases, respiratory system diseases, metabolic and skeletal system diseases, or malignant tumors; ⑦Contraindications for intramuscular injection and blood drawing, such as coagulation disorders, thrombosis or hemorrhagic diseases, or situations requiring continuous use of anticoagulants; ⑧Severe hypertension that cannot be controlled by medication (measured on-site: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
8. History of major surgery within 12 weeks prior to enrollment (as determined by the investigator), or not fully recovered from the surgery, or having plans for major surgery during the anticipated period of the subject's participation in the study;
9. History of long-term alcohol abuse and/or drug abuse;
10. Individual who is currently participating in other research or unregistered product (drugs, vaccines, or devices, etc.) clinical studies, or plan to participate in other clinical studies before the end of this clinical study;
11. Other conditions that may impact the subject's safety or influence the assessment of vaccine response, as determined by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The geometric mean titer (GMT) of Neutralizing Antibodies Against RSV A and RSV B | 30 days after vaccination
  Measured by microneutralization assay.
Geometric Mean Fold Rise (GMFR) for Neutralizing Antibodies Against RSV A and RSV B | 30 days after vaccination
  Change from prevaccination in geometric mean fold rise of Neutralizing antibody titer Against RSV A and RSV B

SECONDARY OUTCOMES:
The GMT of Neutralizing Antibodies Against RSV A and RSV B | 14 days, 3 months, 6 months and 12 months after vaccination after vaccination
  Measured by microneutralization assay.
GMFR for Neutralizing Antibodies Against RSV A and RSV B | 14 days, 3 months, 6 months and 12 months after vaccination
  Change from prevaccination in geometric mean fold rise of Neutralizing antibody titer Against RSV A and RSV B
The geometric mean concentration (GMC) for Pre-fusion Protein Specific Binding Antibodies | 30 days, 3 months, 6 months and 12 months after vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
GMFR for Pre-fusion Protein Specific Binding Antibodies | 30 days, 3 months, 6 months and 12 months after vaccination
  Change from prevaccination in geometric mean fold rise of Pre-fusion Protein Specific Binding Antibodies
Occurrence of immediate adverse events | Within 30 minutes after vaccination
  The incidence and severity of any adverse events (AEs) within 30 minutes after vaccination
Incidence of solicited AE | Within 0-7 days after vaccination
  Occurrence and severity of solicited local injection site reactions for 7 days (Day 0-Day 7) following vaccination. (i.e., pain, redness, swelling).
  Occurrence and severity of solicited systemic reactions for 7 days (Day 0-Day 7) following vaccination. (i.e., myalgia, fatigue, headache, chills, fever).
Incidence of unsolicited AEs | Within 0~30 days after vaccination
  The incidence and severity of any unsolicited AEs, including all AEs, except solicited AEs reported Day 0~30 after the vaccination.
Occurrence of serious adverse events (SAEs) and adverse events of special interests (AESIs) | 12 months after vaccination
  Incidence and severity of Serious adverse events and adverse events of special interest within 12 months after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yeqing Tong, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Center for Disease Control and Prevention of Dangyang City, Dangyang, China

IPD SHARING:
Plan to Share IPD: Undecided